CLINICAL TRIAL: NCT02546882
Title: Phase 1/2 Study of Autologous Stromal Vascular Fraction in Adipose Tissue Transplantation in Improving Skin Grafting
Brief Title: The Improving Effect of Autologous Stromal Vascular Fraction (SVF) in Adipose Tissue on Skin Grafting
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: West China Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Second Affiliated Hospital of Suzhou University (Other); The First People's Hospital of Zhaoqing City (Unknown); Wuhan Third Hospital (Other)
Responsible Party: Principal Investigator, Qing-Feng Li, MD, PhD, Professor, Head of the Department of Plastic and Reconstructive Surgery, Shanghai 9th People'sHospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012BAI11B03; 2012BAI11B03 (Other Grant/Funding Number: Scientific and Technical Supporting Programs)
Record Dates: First submitted 2014-01-23; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Skin; Deformity, Due to Scar
Keywords: stromal vascular fraction; skin graft
MeSH Terms: conditions — Congenital Abnormalities | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- stromal vascular fraction (Experimental): The adipose tissue in abdomen or thigh will be harvested and digested at 37 °C for 60 min with 0.2% collagenase I/Ⅲ. After filtration and centrifugation, mature adipocytes are separated from the cell pellet. The pellet then is treated with erythrocyte lysis buffer twice to remove red cell fragment. The harvested pellet is stromal vascular fraction (SVF).
  Interventions: Biological: stromal vascular fraction
- saline (Placebo Comparator): 1 ml saline without cells will be used as placebo.
  Interventions: Drug: saline

INTERVENTIONS:
Biological: stromal vascular fraction — 1million stromal vascular fraction was resuspended in 1 ml saline and transplanted for 1 cm2 area.
  Other Names: heterogeneous cell populations isolated from adipose tissue
  Arms: stromal vascular fraction
Drug: saline — 1 ml saline was injected for 1 cm2 area.
  Other Names: normal saline
  Arms: saline

SUMMARY:
The purpose of this study is to observe whether the transplantation of autologous stromal vascular fraction (SVF) in adipose tissue is safe and its effect on improving the texture and contracture of skin grafting.

DETAILED DESCRIPTION:
Reconstruction of large scale skin defect is still a challenge for clinical surgeons. The application of skin grafting works as an important choice, however, the strong contracture and poor appearance limit its wide application in scar repair. The stromal vascular fraction (SVF) of adipose tissue is a group of heterogeneous cells including multipotential mesenchymal cells, preadipocytes, endothelial cells, fibroblasts, macrophages and smooth muscle cells. Previous researches have reported that SVF could secrete various angiogenic growth factors in vitro and enhance neovascularisation of ischaemic tissue in vivo. The Adipose-derived Stem cells in the SVF are multipotential stem cells which have the ability to regenerate, while differentiating to become adipose tissue and help to improve the texture of the grafted skin. Besides, SVF is easy to be harvested in large numbers with less donor injury and can be used directly after isolation without in vitro culture, which makes it a good alternative for regenerative medicine.This study is to observe the effect of autologous SVF on improving the texture and contracture of skin grafting.

Patients requiring skin graft of 2 symmetry parts of the body between the age of 3 and 70 years will be enrolled and randomized into two groups, named as the experimental group with SVF transplantation and the control group with no cell transplantation. Patients from the experimental group will have a fat aspiration on the surgery day. The adipose tissue in abdomen or thigh will be digested at 37 °C for 60 min with 0.2% collagenase IV. After filtration and centrifugation, mature adipocytes are separated from the cell pellet. The pellet then is treated with erythrocyte lysis buffer twice to remove red cell fragment. The harvested pellet is SVF. The SVF will be resuspended in saline and transplanted between the grafted skin and the wound with 1 million cells for 1 cm2 area. Skin thickness, texture, contracture and colour will be observed to measure the effect of SVF on skin grafting post treatment.

ELIGIBILITY:
Inclusion Criteria:

* With symmetrical scar or soft tissue deficiencies requiring skin graft therapy.
* Age of 3 to 70.
* Have no underlying disease except skin scar deformity.
* Have enough healthy donor site skin for both sides of receiving area.

Exclusion Criteria:

* Not fit for skin graft treatment;
* Evidence of infection, ischemia, ulcer or other pathological changes within the targeting area which defined as not suitable for skin grafting; or history of delayed healing, radiational therapy;
* Significant renal, cardiovascular, hepatic and psychiatric diseases;
* Significant medical diseases or infection (including but not limited to the carrier of hepatitis B virus or HIV);
* BMI >30;
* Alcohol abuse
* History of any hematological disease, including leukopenia , thrombocytopenia, or thrombocytosis;
* Evidence of malignant diseases or unwillingness to participate.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Measure the texture and colour change of the skin using Cutometer® dual MPA 580 and questionnaires in 6 months post the treatment. | 6 months post the treatment.
  Questionnaires scores satisfaction range from 0(not satisfied with the result) to 10(good result)

SECONDARY OUTCOMES:
Occurence of major adverse events | Up to approximately 18 months after study start
  Including skin graft ischaemia, necrosis, infection, and all other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Qingfeng Li, MD, PhD, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Qin J, Cheng C, Huang RL, He J, Zhou S, Tan PC, Zhang T, Fang B, Li Q, Xie Y. Isolation of the Stromal Vascular Fraction Using a New Protocol with All Clinical-Grade Drugs: From Basic Study to Clinical Application. Aesthetic Plast Surg. 2024 Nov;48(22):4702-4711. doi: 10.1007/s00266-024-04221-9. Epub 2024 Jul 10. PMID 38987318